CLINICAL TRIAL: NCT05692466
Title: Discovering Novel Cancer Treatment Options Using a Comprehensive NGS-based Molecular Testing Panel in the Community Setting ("DINOSAur")
Acronym: DINOSAur
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Glendale Adventist Medical Center d/b/a Adventist Health Glendale (Other)
Collaborators: Caris Life Sciences (Industry)
Responsible Party: Principal Investigator, Mihran Shirinian, Principal Investigator, Glendale Adventist Medical Center d/b/a Adventist Health Glendale
Other Study IDs: DINOSAur
Record Dates: First submitted 2021-12-21; First posted 2023-01-20 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Stage III Solid Tumors; Stage IV Solid Tumors

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Active: Newly diagnosed cancer patients.
  Interventions: Diagnostic Test: Comprehensive molecular panel test; Other: EORTC QLQ-30
- Control: Historically diagnosed cancer patients.

INTERVENTIONS:
Diagnostic Test: Comprehensive molecular panel test — Lab test
  Groups: Active
Other: EORTC QLQ-30 — Quality of life questionnaire
  Groups: Active

SUMMARY:
To prospectively identify cancer patients whose tumors express specific molecular markers targeted by therapeutic agents from a comprehensive molecular test, for the purpose of selecting the most clinically appropriate treatment in a pragmatic two arm trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have given informed consent in accordance with the methods and procedures of this study
* Diagnosis of cancer (stage 3 and stage 4; solid tumors only) requiring medical care
* Patients who have not received treatment related to his/her cancer
* Patients who are willing to sign a release of medical records to the research team
* Male and female patients ≥18 years of age
* Patients under oncology care of a participating site
* Sufficient clinical status for collection of biospecimen samples within usual care
* Patients who have insurance coverage for CMT

Exclusion Criteria:

* Patients considered minors in the jurisdiction where the protocol is conducted.
* Patients who are prisoners and pregnant women.
* Patients who cannot provide consent and did not sign a power of attorney.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed cancer patients at the pathology level.
Sampling Method: Probability Sample
Enrollment: 572 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
European Organization for Research and Treatment of Cancer quality of life Questionnaire-C30 (QLQ-C30) | 2 years
  The EORTC Core Questionnaire (QLQ-C30) includes six clearly distinguishable functioning scales that have been thoroughly tested and validated on an international level and that are available in 110 different language versions.

SECONDARY OUTCOMES:
Compare the proportion of patients enrolling in clinical trials | 2 years
  To compare the proportion of enrolling in clinical trials between cancers patients who received the CMT versus cancer patients with no CMT.

CONTACTS AND LOCATIONS:
Locations (1):
- Adventist Health Glendale, Glendale, California, United States

IPD SHARING:
Plan to Share IPD: No